CLINICAL TRIAL: NCT06653114
Title: Development and Evaluation of an Educational Program for the Management of Chronic Musculoskeletal Pain, With an Emphasis on Pain Neuroscience and the Development of Communication Skills for Physiotherapists
Brief Title: Development and Evaluation of an Educational Program for the Management of Chronic Musculoskeletal Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Konstantina Savvoulidou, PhD Student, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 12
Record Dates: First submitted 2024-10-19; First posted 2024-10-22 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Chronic Musculoskeletal Pain; Clinical Communication
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chronic Musculoskeletal Pain + Communication skills (Experimental): Participants will complete both parts of the educational program (assessment and management of chronic musculoskeletal pain and development of communication skills).
  Interventions: Other: Education in Chronic Musculoskeletal Pain; Other: Education in Communication Skills
- Chronic Musculoskeletal Pain (Experimental): Participants will complete only the management of chronic musculoskeletal pain portion of the educational program.
  Interventions: Other: Education in Communication Skills

INTERVENTIONS:
Other: Education in Chronic Musculoskeletal Pain — Improving Knowledge and Skills in Chronic Musculoskeletal Pain (Assessment and Management)
  Arms: Chronic Musculoskeletal Pain + Communication skills
Other: Education in Communication Skills — Developing Communication Skills (Empathy, Motivational Interviewing, Shared Decision-making)

SUMMARY:
A controlled randomized study will be conducted to assess the effectiveness of the educational program before and after its implementation. An invitation to participate will be extended to physiotherapists interested in the training program. More than 64 physiotherapists will be randomly assigned to two equal groups. All participants will sign an informed consent form before the commencement of the study and will be informed about the study's content, duration, and their right to withdraw at any time. A structured educational program consisting of two parts will be developed, encompassing three core modules (Part A) on the management of chronic pain and three core modules (Part B) on communication skills and techniques. The modules in Part A of the educational program will focus on elucidating the neurophysiological mechanisms of pain, performing differential assessments based on chronic musculoskeletal pain phenotypes, and addressing and managing the factors contributing to patients' pain experiences and rehabilitation, with a particular emphasis on pain neuroscience education. The modules in Part B of the educational program will concentrate on the development of communication skills essential for effective interaction between patients and physiotherapists. The first group will complete all modules of the educational program, while the second group (control group) will only participate in the Part A education modules. The effectiveness of the program will be evaluated before and after its implementation by two independent examiners through the administration of an Objective Structured Clinical Examination (OSCE) and the use of reliable and valid questionnaires and scales.

DETAILED DESCRIPTION:
A controlled randomized study will be conducted to assess the effectiveness of the educational program before and after its implementation. An invitation to participate will be extended to physiotherapists interested in the training program. More than 64 physiotherapists will be randomly assigned to two equal groups. All participants will sign an informed consent form before the commencement of the study and will be informed about the study's content, duration, and their right to withdraw at any time. A structured educational program consisting of two parts will be developed, encompassing three core modules (Part A) on the management of chronic pain and three core modules (Part B) on communication skills and techniques. The modules in Part A of the educational program will focus on elucidating the neurophysiological mechanisms of pain, performing differential assessments based on chronic musculoskeletal pain phenotypes, and addressing and managing the factors contributing to patients' pain experiences and rehabilitation, with a particular emphasis on pain neuroscience education. The modules in Part B of the educational program will concentrate on the development of communication skills essential for effective interaction between patients and physiotherapists. The first group will complete all modules of the educational program, while the second group (control group) will only participate in the Part A education modules. The effectiveness of the program will be evaluated before and after its implementation by two independent examiners through the administration of an Objective Structured Clinical Examination (OSCE) and the use of reliable and valid questionnaires/scales. Upon completion of the program and its evaluation, participants in the control group will have the opportunity to complete the communication skills training as well.

ELIGIBILITY:
Inclusion Criteria:

* Physiotherapists registered with the Panhellenic Association of Physiotherapists
* >2 years of clinical experience with chronic musculoskeletal patients

Exclusion Criteria:

* Participants who have attended any educational program or seminar related to pain education, pain neuroscience education, or a training program related to improving communication skills lasting more than 6 hours

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-10-19 (Actual); Primary Completion 2025-01-11 (Actual); Study Completion 2025-01-11 (Actual)

PRIMARY OUTCOMES:
Change on Baseline in Knowledge on Pain (the Knowledge and Perceptions about Pain (KNAP) Questionnaire at Week 5 and Week 12 | Baseline, Week 5 and Week 16
  The Knowledge and Perceptions about Pain (KNAP) Questionnaire is a 30-item questionnaire. These questions are designed to assess various aspects of pain knowledge and beliefs, including the understanding of pain mechanisms, treatment approaches, and the impact of pain on individuals. It uses a Likert Scale (1 strongly disagree - 6 strongly agree). A higher KNAP score indicates that an individual's knowledge and attitudes about pain align more closely with current pain neuroscience.
Change on Baseline in Knowledge on Pain (The Revised Neurophysiology of Pain Questionnaire (R-NPQ) at Week 5 and Week 12 | Baseline, Week 5 and Week 16
  The revised Neurophysiology of Pain Questionnaire (R-NPQ) developed to assess knowledge about the biological and physiological mechanisms of pain. Created by Dr. Lorimer Moseley in 2003 and revised by Ostelo et al. 2013. It evaluates understanding of how the nervous system and brain process pain. The total score is the sum of points from all correctly answered questions.
Change on Baseline in Empathy (The Toronto Components Empathy Questionnaire (ECQ) at Week 5 and Week 12 | Baseline, Week 5 and Week 16
  The Toronto Components Empathy Questionnaire (ECQ) is designed to assess different aspects of empathy, particularly in clinical settings (Spreng et al., 2009). Developed to measure how individuals perceive and respond to others' emotions. 26 items are allocated for professional life, with an equal distribution between cognitive and emotional empathy.
Change on Baseline in using of Share Decision-Making (Shared Decision-Making Questionnaire (SDM-Q-9) at Week 5 and Week 12 | Baseline, Week 5 and Week 16
  The SDM-Q-9 is a validated 9-item questionnaire designed to evaluate patients' perceptions of shared decision-making (SDM) (Kriston et al., 2010). Each item represents a distinct step in the SDM process and is rated on a 6-point Likert scale from 0 ("completely disagree") to 5 ("completely agree").
Change on Baseline in communication and clinical skills using an objective structured clinical examination (OSCE) at Week 5 and Week 12 | Baseline, Week 5 and Week 16
  The Objective Structured Clinical Examination (OSCE) is a comprehensive and structured assessment to evaluate clinical skills and competencies in healthcare professionals. OSCE will be used to assess the following focused clinical skills of participants: history taking, gathering information, information provided in patients, empathy, share decision-making, motivational interviewing.

CONTACTS AND LOCATIONS:
Overall Officials: Eleni V Kapreli, Prof, Study Director — University of Thessaly
Locations (1):
- University of Thessaly, Lamia, Greece